CLINICAL TRIAL: NCT05324514
Title: Full-Thickness Microscopic Skin Tissue Column Grafting Technique Using the ART (Autologous Regeneration Tissue) System: An Interventional Clinical Trial
Brief Title: Microscopic Skin Tissue Column Grafting Technique Using the Autologous Regeneration of Tissue System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ART-1
Record Dates: First submitted 2019-10-03; First posted 2022-04-12 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Wound of Skin; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Participants will have three wound sites that will be randomized to receive either the standard of care treatment, high density microscopic tissue skin columns, or low density microscopic tissue skin columns.
Who Masked: Outcomes Assessor
Masking Description: Formalin embedded biopsies will be sectioned and the sections will be stained. Stained tissue sections will be graded by blinded dermato-pathologists.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Standard of Care (Active Comparator): STSG grafting application.
  Interventions: Procedure: Split-thickness skin grafting
- High Density (Experimental): MSTC high density application.
  Interventions: Device: High density microscopic skin tissue column grafting
- Low Density (Experimental): MSTC low density application.
  Interventions: Device: Low density microscopic skin tissue column grafting

INTERVENTIONS:
Procedure: Split-thickness skin grafting — Harvesting for split-thickness skin grafting will be performed at the specified donor site using a pneumatically powered dermatome with a setting of 10 /1000th inch and meshed 2:1.
  Arms: Standard of Care
Device: High density microscopic skin tissue column grafting — MSTC harvest will be conducted using the ART system (Medline Industries) in accordance with the manufacturer's instructions and distributed at high density (300-360 columns/50cm2).
  Arms: High Density
Device: Low density microscopic skin tissue column grafting — MSTC harvest will be conducted using the ART system (Medline Industries) in accordance with the manufacturer's instructions and distributed at low density (150-180 columns/50cm2).
  Arms: Low Density

SUMMARY:
This study evaluates Microscopic Skin Tissue Column (MSTC) grafting technique using the Autologous Regeneration Tissue (ART) System in the treatment of skin loss. Each participant will have three study treated areas, the three treatments include: 1. traditional grafting, 2. high density MSTC, 3. low density MSTC.

DETAILED DESCRIPTION:
The current standard of care for coverage of large open wounds is split-thickness skin graft (STSG). These STSGs are typically harvested with a dermatome, which tangentially removes the epidermis and a thin layer of dermis from a healthy donor site. While relatively versatile, there are important limitations to STSGs. First, a healthy and readily accessible donor site is required prior to grafting. Second, each donor site itself becomes an open wound and is unable for grafting for approximately two weeks as the wound heals. To facilitate wound coverage, harvested STSG can be meshed up to a rate of 6:1 (though more common ratios are 1:1 and 2:1). However, widely meshed grafts tend to produce more severe scars and contractures, which represent tremendous long-term morbidity to the patient.

The only means to avoid using widely meshed grafts is to harvest additional healthy donor skin, resulting in more pain from larger wound burdens and disfiguring scars in previously uninjured regions. Finally, STSG does not include deeper dermal structures such as hair follicles and sweat glands, and as such these grafts are both functionally and aesthetically substandard. Recently, skin microcolumn grafting has been proposed to address both skin graft donor site morbidity and long-term graft contracture. Specifically, the Autologous Regeneration of Tissue (ART)TM System, an FDA-cleared device, harvests full-thickness microscopic skin tissue columns (MSTC) orthogonally instead of tangentially; each skin column includes epidermis, dermis and associated adnexal structures, and subcutaneous fat. These MSTC cover an area up to 10x larger than the donor site (100:1 ratio, compared to up to 6:1 using STSG). Inclusion of adnexal structures results in improved wound-healing quality, less scarring, and a lower rate of secondary contracture. The small wounds caused by the ART system at the donor site during MSTC harvesting heal quickly and without the comorbidities associated with traditional harvesting. This autologous approach maintains low immunogenicity as no foreign or synthetic tissue is used as a skin substitute, which decreases the chance of infection or rejection in the wound bed. In short, the ART system allows for expansion of a donor site to a ratio of 1:100, faster healing of the donor site while still preserving donor site function, and improved healing of the original wound.

The investigators will conduct a prospective, randomized controlled clinical trial comparing the MSTC grafting technique to the standard of care. Treatment sites will be randomized to either receiving MSTC or the traditional STSG. Objective measurements and assessments will be completed during subject follow-ups visits for up to six months.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 and age less than or equal to 70.
* Skin loss from surgery, trauma, and/or burns.
* Presence of one uniform contiguous wound ≥150cm2
* Sufficient non-injured healthy skin from which conventional STSG can be harvested to cover study and non-study sites.
* Sufficient non-injured healthy skin from which the study device can be used to harvest MSTC to cover the study sites.
* Study donor site has not been previously harvested.
* Able and likely to follow-up, to have three consecutive appointments and appear for 6 month follow up visit.
* Subject agrees to abstain from enrollment in any other interventional clinical trial while enrolled in this study.

Exclusion Criteria:

* Exposure of tendon, bone devoid of peritenon or periosteum, or other structures deemed non-graftable by the treating physician or study investigator.
* Concomitant skin disease/infection at the recipient or donor sites.
* Use of topical steroid, anti-metabolite, or other pharmacologic therapy on study site.
* Use of systemic steroids in the past month.
* Concurrent conditions that in the opinion of the investigator may compromise subject safety, study objectives or wound healing.
* Current recipient of immunosuppressive therapy.
* Current treatment with medication that inhibit/compromise wound healing.
* Known history of malignancy.
* Pregnancy or lactation
* Prisoner
* History of noncompliance ->40% total body surface area involvement.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of healing | Day 7
  The rate of healing of the donor sites will be assessed utilizing clinical assessments and photography with 3D camera and the Silhouette Star wound camera.
Rate of epithelialization | Day 7
  The rate of epithelialization will be assessed utilizing clinical assessments and photography with 3D camera and the Silhouette Star wound camera.
Rate of healing | Day 14
  The rate of healing of the donor sites will be assessed utilizing clinical assessments and photography with 3D camera and the Silhouette Star wound camera.
Rate of epithelialization | Day 14
  The rate of epithelialization will be assessed utilizing clinical assessments and photography with 3D camera and the Silhouette Star wound camera.

SECONDARY OUTCOMES:
Incidence of pain | Day 3- Month 6
  Donor sites will be assessed for incidence and level of pain experienced.
Skin function | Day 17- Month 6
  Skin function as measures by the validated Patient and Observer Scar Assessment Scale. The Patient and Observer Scar Assessment scale uses a 0-10 scale 0 being normal appearance, 10 being the worst possible outcome (POSAS).
Presence of adnexal structures | Day 30, Month 6
  Presence of adnexal structures will be assessed by obtaining a wound biopsy.
Reepithelization | Day 3- month 6
  Clinical assessment for the need to re-graft treatment sites.
Skin appearence | Day 17- Month 6
  Skin appearance measured using Vancouver Scar Scale (VSS). VSS rates Vascularity, pigmentation, pliability, and hight of the affected skin using a numeric scale to get an overall total of 1-13.
Skin pliability | Day 17- Month 6
  Skin pliability measured using a Dermal torque meter (DTM).
Skin integrity | Day 17- Month 6
  Skin integrity measured by a tewameter. The tewameter is a measuring device for the assessment of the trans-epidermal water loss (TEWL).
Skin pressure | Day 17- Month 6
  Skin pressure measured using a semmes-weinstein aesthesiometer
Skin color | Day 17- Month 6
  Skin color to be measured using colorimeter.

IPD SHARING:
Plan to Share IPD: No